CLINICAL TRIAL: NCT07132957
Title: A Phase I Study to Evaluate the Mass Balance of 14C-labeled AL8326 in Healthy Subjects
Brief Title: A Study of AL8326 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Advenchen Laboratories Nanjing Ltd. (Industry)
Responsible Party: Sponsor
Organization: Advenchen Laboratories, LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AL8326-CN-011
Record Dates: First submitted 2025-02-19; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Small Cell Lung Cancer; Solid Tumors
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 14C-labeled AL8326 (Experimental): Single dose
  Interventions: Drug: 14C-labeled AL8326

INTERVENTIONS:
Drug: 14C-labeled AL8326 — Oral, About 60mg (200μCi) of 14C-labeled AL8326

SUMMARY:
This experiment plans to enroll 6-8 healthy male subjects in China, and ultimately collect complete test samples and data from at least 6 subjects as the standard. On the first day of the experiment, each subject orally took a single dose of [14C] AL8326 oral formulation containing approximately 60mg (200 μ Ci). During the experiment, whole blood, plasma, urine, and fecal samples were collected at designated time points/time periods.

DETAILED DESCRIPTION:
This experiment adopts a single center, open label, non randomized, single dose trial design. By measuring the total radioactivity, calculate the ratio of total radioactivity in whole blood to plasma of [14C] AL8326, pharmacokinetic parameters, recovery rate, and excretion pathway data of total radioactivity in plasma. At the same time, by identifying the spectra of radioactive metabolites and the structures of major metabolites in plasma, urine, and feces, the main metabolic elimination pathways and characteristics of AL8326 in the human body were obtained, as well as the circulating metabolites that are close to or higher than 10% of the total radioactive exposure in plasma.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for this study:

1. Chinese healthy male subjects, 18 to 45 years of age (inclusive)
2. Body mass index (BMI) of 19-26 kg/m2 (inclusive), and body weight not less than 50 kg (inclusive)
3. Subjects who had no fertility or sperm donation plan from signing the informed consent until 1 year after the end of the trial, or those who agreed that the subjects and their partners should strictly use contraception from signing the informed consent until 1 year after the end of the trial; Voluntarily signing the ICF，Ability to communicate well with the investigator and compliance to complete the trial according to the protocol.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Clinically significant abnormality of physical examination, vital signs, routine laboratory tests (hematology, blood chemistry, coagulation, urinalysis, and stool routine + occult blood), 12-lead ECG, chest X-ray (anterograde), digital anal examination, thyroid function,ophthalmic examination and abdomen ultrasound (liver, gallbladder, pancreas, spleen, and kidneys), etc.
2. Subjects with an allergic constitution, such as known allergic history to two or more substances, or allergic diseases, or those who may be hypersensitive to the investigational drug or its excipients, as judged by the investigator;
3. Gastrointestinal diseases causing clinically significant symptoms such as nausea, vomiting, diarrhea, or malabsorption syndrome; Or a history of severe vomiting or diarrhea within one week before the screening period;
4. History of dysphagia or any condition that may affect drug absorption (e.g., gastrectomy, cholecystectomy, gastric bypass, duodenotomy, colectomy);
5. History of any clinical critical illness or presence of diseases or conditions that the investigator considers may affect the trial results, including but not limited to diseases of digestive system, circulatory system, respiratory system, endocrine system, nervous system, urinary system or blood, immune system, psychiatric system and metabolism and nutrition diseases ;
6. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, torssion ventricular tachycardia, ventricular tachycardia, long QT syndrome or family history (genetic proof or sudden death of a close relative at a young age);
7. Major surgery within 6 months before screening or incomplete healing of surgical incision, the major surgeries including but not limited to any procedures that have significant risk of hemorrhage, prolonged general anesthesia, open biopsy, or marked traumatic invasive injury;
8. History of active bleeding (e.g., peptic ulcer, intracranial hemorrhage, skin ecchymosis, gingival bleeding); History of any disease within the previous 6 months that may increase the risk of bleeding (such as tumor bleeding, spontaneous hematoma, eye bleeding, hemoptysis, gastrointestinal bleeding or ulcers,hematuria,reproductive system bleeding, traumatic hematoma/bleeding, and frequent epistaxis/gingival bleeding/subcutaneous or skin bleeding) were screened.
9. Hemorrhoids or perianal diseases with regular/current hematochezia;
10. Hepatitis B surface antigen , hepatitis C virus antibody IgG test, human immunodeficiency virus antigen/antibody combination test, or Treponema pallidum antibody test is positive
11. Use of any drug that affects drug metabolism enzymes or transporters (P-gp and BCRP) in the 30 days prior to screening, as detailed in Appendix 5;
12. Have taken any prescription drugs, over-the-counter drugs, Chinese herbs or food supplements (vitamins, calcium supplements) in the 14 days prior to screening and before dosing;
13. Participation in any other clinical trial (including drug and device clinical trials) within 3 months before screening;
14. Habitual constipation or diarrhea;
15. History of blood loss or donation (≥400mL) within 3 months before screening, received a transfusion or blood component within 1 month, or planned to donate blood within 3 months after the end of the trial;
16. Daily smoking exceeding 5 cigarettes (≥ 5 cigarettes) within 3 months before Screening, or habitual use of nicotine-containing products and inability to withdraw during the trial period;
17. Alcoholism or frequent alcohol use within 6 months before screening, i.e., weekly alcohol consumption > 14 units (1 unit = 360 mL of beer or 45 mL of ABV 40% spirit or 150 mL of wine),Or alcohol breath test >20mg/dL，or unable to abstain during the test
18. Drug abuse, use of soft drug (e.g., marijuana) within 3 months before screening, or use of hard drug (e.g., cocaine, amphetamines, phencyclidine, etc.) within 1 year before screening; or positive urine drug test at screening;
19. Habitual or excessive (more than 8 cups a day, 1 cup =250mL) consumption of grapefruit juice, tea, coffee and/or caffeinated beverages, and unable to abstain during the trial period;
20. Those who have special requirements for diet and cannot abide by the uniform diet;
21. History of long-term exposure to radioactive conditions, or significant radiation exposure (≥2 chest/abdominal CT, or ≥3 other kinds of X-ray examinations) within 1 year before administration, or participating in radiopharyngology labeling tests;
22. History of needle fainting and blood fainting, difficulty in blood collection or inability to tolerate venous puncture blood collection;
23. Vaccinated within 1 month before screening or planned to be vaccinated during the trial period;
24. Subjects who with poor adherence or have any factors that make them not suitable for participating in this trial, as assessed by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Material balance | All excreted urine and feces samples at specified time points during 0-480 hours after dosing will be collected.
  the cumulative excretion rate of total radioactive material in excreta (urine and feces);
Metabolites | Conduct testing within 1 month after all subjects collect plasma, urine, and fecal samplesat all time points required by the protocol
  The percentage of the original drug and each metabolite in urine and feces (% dose)
Metabolites | Conduct testing within 1 month after all subjects collect plasma samplesat all time points required by the protocol
  The AUC percentage of the original drug and circulating metabolites in plasma (%AUC) were calculated;
Pharmacokinetic | Conduct testing within 1 month after all subjects collect plasma samplesat all time points required by the protocol
  Pharmacokinetic parameters for total radioactivity in plasma， including peak concentration (Cmax), time to peak (Tmax), area under the drug-time curve (AUC0-t and AUC0-∞), elimination half-life (t1/2), apparent clearance (CL/F), apparent volume of distribution (Vd/F) and mean residence time (MRT). ) and mean residence time (MRT).
whole blood | Conduct testing within 1 month after all subjects collect plasma samplesat all time points required by the protocol
  whole blood to plasma total radioactivity partition ratio

SECONDARY OUTCOMES:
Plasma pharmacokinetics | Conduct testing within 1 month after all subjects collect plasma, urine, and fecal samplesat all time points required by the protocol
  PK parameters of AL8326 and its main metabolites in plasma， including peak concentration (Cmax), time to peak (Tmax), area under the drug-time curve (AUC0-t and AUC0-∞), elimination half-life (t1/2), apparent clearance (CL/F), apparent volume of distribution (Vd/F) and mean residence time (MRT). ) and mean residence time (MRT).
Safety | From signing the ICF until 22 days after the first dosing
  Number of participants with adverse events/drug-related adverse events, with abnormal physical examination findings, abnormal vital signs, abnormal 12-lead electrocardiogram, and abnormal laboratory tests results

CONTACTS AND LOCATIONS:
Overall Officials: LiYan Miao, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No